CLINICAL TRIAL: NCT03222297
Title: Effects of Early Skull Repair With Titanium Mesh on Cerebral Blood Flow and Neurological Recovery: a Randomized Controlled Clinical Trial Based on CT Perfusion Evaluation
Brief Title: Effects of Early Skull Repair With Titanium Mesh on Cerebral Blood Flow and Neurological Recovery
Status: Completed | Type: Observational
Sponsor: Taihe Hospital (Other)
Responsible Party: Principal Investigator, Yase Zhuang, Principal Investigator, Taihe Hospital
Other Study IDs: TaiheH_002
Record Dates: First submitted 2017-07-12; First posted 2017-07-19 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- test group: Patients with craniocerebral injury were randomized into test group (n = 40) with early skull repair using titanium mesh within 1-3 months after decompression.
  Interventions: Device: early skull repair
- control group: Patients with craniocerebral injury were randomized into control group (n = 46) with late-stage skull repair using titanium mesh within 6-12 months after decompression.
  Interventions: Device: late-stage skull repair

INTERVENTIONS:
Device: early skull repair — Patients with craniocerebral injury were randomized into test group (n = 40) with early skull repair using titanium mesh within 1-3 months after decompression.
  Other Names: test group
  Groups: test group
Device: late-stage skull repair — Patients with craniocerebral injury were randomized into control group (n = 46) with late-stage skull repair using titanium mesh within 6-12 months after decompression.
  Other Names: control group
  Groups: control group

SUMMARY:
To evaluate the feasibility of CT perfusion technique to monitor the changes of blood perfusion in the brain tissue before and after skull repair using titanium mesh. To determine the best timing for skull repair using the three-dimensional titanium mesh; to compare the effects of early (1-3 months after decompression) and late-stage (6-12 months after decompression) skull repair on neurologic rehabilitation.

DETAILED DESCRIPTION:
A skull defect is inevitable in patients with traumatic brain injury undergoing decompression treatment, which results in a loss of physiological and functional integrity of the brain that makes atmospheric pressure directly act on the brain tissue to induce environmental disorders in the brain. Moreover, with the changes in the body position, the contents of the brain often move in an unstable position, and with the extension of time, there may be compensatory ventricular enlargement and brain atrophy, eventually causing neurological dysfunction and cognitive disorders. Therefore, it is imperative to repair the skull defect.

There are many repair materials for skull defects, including autogenous bone, allogeneic bone, nonmetallic materials (plexiglass, bone cement, silicone rubber, etc.) and titanium mesh. The performance of different materials have their own advantages and disadvantages, and titanium alloy is an ideal repair material and has been widely used in clinical practice because of good biocompatibility and strength, no aging, low density, non-iron atoms, ability to be not magnetized in magnetic fields, and no influence on CT, MRI, EEG and X-ray examination.

The timing for repair of skull defect after traumatic brain injury is still controversial. Some scholars believe that if there is no hydrocephalus and intracranial infection after decompression with removal of bone flap, skull repair should be proceeded as soon as possible to isolate the scalp from the dura mater and recover the normal intracranial pressure by easing the negative effects of the scalp, such as cerebrovascular traction, compression and distortions. Most importantly, early skull repair is able to reduce a variety of secondary neurological deficits due to skull defects, increase brain surface blood flow, and thus reduce epileptic attack. Of course, some scholars recommend late-stage skull repair, and they believe hematoma absorption after decompressive surgery is a long process, and in some patients, hematoma will be completely absorbed in about 3 months or even longer, which may result in secondary brain edema. Moreover, surgical trauma exerts negative effect on the brain tissue recovery, which is not conducive to neurologic rehabilitation.

As there is no unified conclusion on the timing for the repair of skull defects, investigators conducted a multi-sample, double-blind, randomized, clinical trial, to collect craniocerebral injury patients undergoing decompression with removal of bone graft who were randomized into two groups to receive early skull repair in test group and late-stage skull repair in control group. CT perfusion technology was used to monitor the blood perfusion in the brain before and after skull repair and to compare the changes of blood perfusion in the brain tissue and neurological recovery in patients undergoing early or late-stage skull repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent decompression via removal of bone flap in the unilateral frontal temporal lobe due to craniocerebral injury and developed no postoperative infection.
* Patients agreed to receive skull repair using titanium mesh.
* Patients and their families agreed to receive CT perfusion examination.
* Patients and their families fully understood the study protocol and agreed to participate in the trial, and then singed the informed consent before the trial.

Exclusion Criteria:

* Hypertension and diabetes out of control, severe heart disease, brain tumors, brain abscess, and cerebral infarction
* Diseases that have interfered with localized perfusion data, such as intracranial aneurysms, arteriovenous malformations
* Combined with depressed skull fractures and skull base fractures
* Hydrocephalus

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eighty-six patients with craniocerebral injury who had undergone decompression with removal of bone flap from January 2013 to January 2016 were recruited and subjected to skull repair using titanium mesh. All the patients were randomized into two groups: test group (n = 40) with early skull repair within 1-3 months after decompression and control group (n = 46) with late-stage skull repair within 6-12 months after decompression.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
blood perfusion in the brain tissue | changes from day 3 before surgery to day 10 after surgery
  To monitor the changes of blood perfusion in the brain tissue based on CT perfusion technology after skull repair with titanium mesh. 50 mL of iopromide was injected at a rate of 5 mL/s into the median cubital vein of the patients, and 3 seconds later, 256-slice spiral CT (Philips) was used for continuous scan for 50 seconds, followed by image processing using a Philips-specific workstation.

SECONDARY OUTCOMES:
Barthel index | at day 30 after surgery
  To measure performance in activities of daily living. The full scores of Barthel index is 100. A higher score is associated with a greater likelihood of being able to live: > 60, mild disability with the ability to basically take care of oneself; 40-60, moderate disability with the need for help in activities of daily living; 20-40, severe disability with the need for great help in activities of daily living; < 20, complete disability with the inability to care for oneself.

IPD SHARING:
Plan to Share IPD: Undecided